CLINICAL TRIAL: NCT02262143
Title: Efficacy and Safety of Combination Therapy of Rosuvastatin and Fenofibrate Versus Rosuvastatin Monotherapy in Mixed Dyslipidemia Patients
Brief Title: Phase III Study of Rosuvastatin and Fenofibrate Versus Rosuvastatin in Mixed Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-ROFE-301
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Mixed Dyslipidemias
MeSH Terms: interventions — Rosuvastatin Calcium; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Rosuvastatin 10 mg, Fenofibrate 160 mg
  Interventions: Drug: Rosuvastatin; Drug: Fenofibrate
- Comparator (Active Comparator): Rosuvastatin 10 mg
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 10 mg, qd, po
  Other Names: Crestor Tab.
Drug: Fenofibrate — Fenofibrate 160mg, qd, po
  Other Names: Lipidil supra Tab.
  Arms: Experimental

SUMMARY:
Efficacy and safety of combination therapy of rosuvastatin and fenofibrate versus rosuvastatin monotherapy in mixed dyslipidemia patients: A randomized, multi-center, double-blind, phase 3 study

ELIGIBILITY:
Inclusion Criteria:

* 19 ~ 80 years old
* High risk patient to Coronary Heart Disease
* At Visit 1(Screening)

  1. Treated with Rosuvastatin 10mg monotherapy 4weeks prior to this study
  2. 110 mg/dl ≥ LDL-C, 200 mg/dl ≤ TG ≤ 500 mg/dl
* At Visit 2 (Baseline), 110 mg/dl ≥ LDL-C, 200 mg/dl ≤ TG ≤ 500 mg/dl

Exclusion Criteria:

* AST or ALT > 2X ULN
* Patients with uncontrolled hyperthyroidism (TSH>1.5X ULN)
* Patients with uncontrolled diabetes (HbA1c ≥ 9%)
* Patients with uncontrolled hypertension(SBP>160mmHg or DBP>95mmHg)
* Patients with congestive heart failure(NYHA class III~IV) or uncontrolled arrhythmia within 6 months
* Patients treated with any investigational drugs within 3 months at the time consents are obtained
* Not eligible to participate for the study at the discretion of investigator

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The mean percent change of Non-HDL Cholesterol | from baseline at week 8

SECONDARY OUTCOMES:
The mean change, percent change of Non-LDL-C | from baseline at week 4
The mean change of Non-LDL-C | from baseline at week 8
The mean percent change of LDL-C, HDL-C, VLDL-C, TG, TC, Apo-AI, Apo-B | from baseline at week 4, 8
The achievement rate of Non-HDL-C<130mg/dl | from baseline at week 4, 8

CONTACTS AND LOCATIONS:
Overall Officials: Jeongtaeck Woo, M.D., Ph.D, Principal Investigator — Kyunghee University Medical Center
Locations (1):
- Ildong Pharm., Seoul, South Korea